CLINICAL TRIAL: NCT01088373
Title: A Phase II Study of the Efficacy and Safety of Lenalidomide Combined to Azacitidine in Intermediate-2 or High Risk MDS With Del 5q
Brief Title: Lenalidomide Combined to Azacitidine in Intermediate-2 or High Risk MDS With Del 5q
Acronym: GFM-AZA-REV-09
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZA-REV-09
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azacitidine, Lenalidomide (Experimental)
  Interventions: Drug: Azacitidine combined to Lenalidomide

INTERVENTIONS:
Drug: Azacitidine combined to Lenalidomide — Azacitidine: 75mg/m2/d for 5 days per cycle of 28 days. Lenalidomide: 5mg/day during 14 days for cohort 1. Lenalidomide: 5mg/day during 21 days for cohort 2. Lenalidomide: 10mg/day during 21 days for cohort 3.
  Other Names: Vidaza.; Revlimid.

SUMMARY:
Higher risk MDS with del(5q) carry very poor prognosis, but show some response to azacitidine and Lenalidomide as single agents . The combination of Lenalidomide and Azacytidine is currently tested in non del 5q MDS patients. Preliminary results have been recently presented at ASH meeting (Sekeres et al, 2007).

Overall, the combination of Lenalidomide and Azacitidine is well-tolerated and early results suggest some efficacy in advanced MDS without del 5q.

In this trial, we will combine Lenalidomide to Azacytidine in higher risk MDS with del (5q).

Patients will receive azacitidine( 75mg/m2/day for 5 days every 28 days) combined to escalating doses of lenalidomide (starting at relatively low dose).

For patients in hematological CR, PR, HI or marrow CR after cycle 2 or 4, it is mandatory to continue on Azacitidine + Lenalidomide as long as there is no unacceptable toxicity or overt progression, with the schedule that yielded response.

In patient still responding after 52 weeks, the drug will continue to be supplied, and follow up until death will be continued in all patients.

ELIGIBILITY:
Inclusion Criteria:

1. age > ou = 18 years and < 75 years.
2. must understand and voluntarily sign an informed consent form.
3. patient considered ineligible for intensive chemotherapy due to age, cardiac contraindication to anthracyclines, comorbidities, previous failure of intensive chemotherapy, or patient willing to avoid intensive chemotherapy.
4. must be able to adhere to the study visit schedule and other protocol requirements.
5. prior thalidomide allowed.
6. documented diagnosis of MDS (according to FAB definition, ie. with marrow blasts up to 30%, or CMML with WBC < 13000/mm3 that meets IPSS criteria for intermediate-2 or high-risk disease.
7. with an associated del 5q[31](the deleted chromosomal region must include 5q[31]), with or without additional cytogenetic abnormalities.
8. female subjects of childbearing potential must:

   * understand the study drug is expected to have a teratogenic risk.
   * agree to have a medically supervised pregnancy test with a minimum sensitivity of 25mIU/ml on the day of the study visit or in the 3 days prior to the study visit once the subject has been on effective contraception for at least weeks. This requirement also applies to women of childbearing potential who practice complete and continued abstinence. the test should ensure the subject is not pregnant when she starts treatment.
   * agree to have a medically supervised pregnancy test every 4 weeks including 4 weeks after the end of study treatment, except in the case of confirmed tubal sterilization. these pregnancy tests should be performed on the day of the study visit or in the 3 days prior to the study visit.

   this requirement also applies to women of childbearing potential who practice complete and continued abstinence.

   * agree to use, and to be able to comply with effective contraception without interruption, 4 weeks before starting study drug throughout the entire duration study drug therapy(including doses interruptions)and for 3 months after the end of the study drug therapy even if she has amenorrhea this applies unless the subject commits to absolute and continuous abstinence confirmed on a monthly basis, to avoid pregnancy for the duration of study.

   the following are effective methods of contraception:
   * implant
   * levonorgestrel-releasing intrauterine system(IUS)
   * Medroxyprogesterone acetate depot, tubal sterilization.
   * sexual intercourse with a vasectomised male partner only(vasectomised must be confirmed by two negative semen analyses), ovulation inhibitory progesterone-only pills(i.e.desogestrel).

   if not established on effective contraception, the female subject must be referred to an appropriately trained health care professional for contraceptive advice in order that contraception can be initiated.

   Because of the increased risk of venous thromboembolism in patients with multiple myeloma taking lenalidomide and dexamethasone, combined oral contraceptive pills are not recommended. If a female subject is currently using combined oral contraception, the patient should switch to one of the effective methods listed above. The risk of venous thromboembolism continues for 4 to 6 weeks after discontinuing combined oral contraception. The efficacy of contraceptive steroids may be reduced during co-treatment with dexamethasone.

   Implants and levonorgestrel-releasing intrauterine systems are associated with an increased risk of infection at the time of insertion and irregular vaginal bleeding. Prophylactic antibiotics should be considered particularly in patients with neutropenia .

   Copper-releasing intrauterine devices are generally not recommended due to the potential risks of infection at the time of insertion and menstrual blood loss which may compromise patients with neutropenia or thrombocytopenia.
   * Understand that even if she has amenorrhea, she must follow all the advice on effective contraception.
   * She understands the potential consequences of pregnancy and the need to rapidly consult if there is a risk of pregnancy
9. Male patients must :

   * Agree the need for the use of a condom if engaged in sexual activity with a woman of childbearing potential. during the entire period of treatment, even if disruption of treatment and during 3 months after end of treatment
   * Agree not to conceive during treatment and study drug therapy (including doses interruptions) and for 3 months after the end of the study drug therapy
   * Agree not to donate semen during study drug therapy and for one week after end of study drug therapy.
   * Agree to learn about the procedures for preservation of sperm., before starting treatment
10. All subjects must :

    * Agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy.
    * Agree not to share study medication with another person and to return all unused study drug to the investigator.
11. Signed informed consent prior to start of any study-specific procedures,
12. Ability to participate to a clinical trial and adhere to study procedures.

    * Criteria for women of non-childbearing potential :

A female patient or a female partner of a male patient is considered to have childbearing potential unless she meets at least one of the following criteria:

* Age ≥ 50 years and naturally amenorrhoeic for ≥ 1 year (amenorrhoea following cancer therapy does not rule out childbearing potential)
* Premature ovarian failure confirmed by a specialist gynaecologist
* Previous bilateral salpingo-oophorectomy, or hysterectomy
* XY genotype, Turner syndrome, uterine agenesis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-03-25 (Actual); Primary Completion 2016-07-25 (Actual); Study Completion 2016-07-25 (Actual)

PRIMARY OUTCOMES:
To identify the "safe most successful dose"(sMSD) that is the dose level where the probabilities of success is maximized across the dose levels and the toxicity rate is kept within acceptable boundaries. | 2 and 4 months of treatment
  Briefly, dose limiting toxicity would be defined by having greater than 30% occurrence of unexpected grade III-IV hematological or non hematological toxicity. Efficacy would be defined as a response rate of 40% after 2 cycles. Overall, 49 patients will be included.

SECONDARY OUTCOMES:
response rate and safety | 36 months
  1. response rate (according to IWG 2006 criteria) to the combination of lenalidomide and azacitidine in adult high and int 2 MDS with del 5q
  2. safety (particularly hematological toxicity) of the combination of Lenalidomide and azacitidine in int-2 and high risk MDS with del 5q [31].
  3. duration of response,
  4. progression to AML,
  5. and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Lionel ADES, MD, Principal Investigator — GFM
Locations (34):
- France (34):
  - Hôpital kremlin Bicêtre, Le Kremlin-Bicêtre, IDF
  - Chu Brabois, Nancy, Vandoeuvre
  - CHU d'Amiens, Amiens
  - CHU Angers, Angers
  - Hôpital de la cote basque, Bayonne
  - Hôpital Avicenne, Bobigny
  - CHU Haut-Lévèque, Bordeaux
  - CH René Dubos, Cergy-Pontoise
  - CHU de, Clermont-Ferrand
  - Centre Hospitalier Sud-Francilien, Corbeil-Essonnes
  - CHU Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - CH Le mans, Le Mans
  - Centre Hospitalier de Lens, Lens
  - CHRU de Limoges, Limoges
  - Hôpital Edouard Heriot, dpt Hématologie Clinique, Lyon
  - Institut Paoli-Calmette, Département d'hématologie, Marseille
  - Centre Hospitalier de Meaux, Meaux
  - Hopital de l'Hotel Dieu, Hematology Dpt, Nantes
  - CHU Archet, Nice
  - CHR La Source orléans, Orléans
  - Hôpital Saint Louis, Paris
  - Saint-Louis Hospital, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital la pitié-Salpétrière, Paris
  - Hopital Cochin Service d'Hématologie, Paris
  - Hôpital Maréchal Joffre, Perpignan
  - Hôpital Jean-Bernard, Poitiers
  - centre hospitalier Jacques Puel, Rodez
  - Hôpital Henri Becquerel, Rouen
  - Hôpital Purpan, médecine Interne, Toulouse
  - Hôpital PURPAN, Service d'Hématologie Clinique, Toulouse
  - CHU Bretonneau, Tours
  - Institut gustave Roussy, Villejuif

REFERENCES:
- See also: Website of the Groupe Francophone des Myélodysplasies (GFM) — http://www.gfmgroup.org/